CLINICAL TRIAL: NCT06157840
Title: Development of an mHealth Behavioral Sleep Medicine Intervention for Use During Medication Assisted Treatment for Opioid Use Disorder
Brief Title: Development of an mHealth Behavioral Sleep Medicine Intervention for Use During Medication Assisted Treatment for MOUD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Allison Wilkerson, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro128158; 1R34DA058511 (NIH)
Record Dates: First submitted 2023-11-06; First posted 2023-12-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use Disorder; Poor Quality Sleep
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth application (Experimental): Study participants, while being stabilized on buprenorphine, will download and engage with the developed mHealth application, completing daily electronic sleep diaries for the next 6 weeks. Each week, they will be asked to complete a short assessment of their experiences from the previous week and their current insomnia severity.
  Interventions: Device: mHealth application and sleep health education
- Control Group (Experimental): Participants in the control group will receive a simplified version of the app with sleep hygiene (SH) instructions and will be required to complete daily electronic sleep diaries for the next 6 weeks. The SH condition will utilize the same application and entail the same daily and weekly logs, but with the didactic material replaced by detailed education about SH strategies. Each week, participants will be asked to complete a brief assessment of their experiences from the previous week and their current insomnia severity.
  Interventions: Device: Simplified mHealth application and sleep health education

INTERVENTIONS:
Device: mHealth application and sleep health education — Study participants will download the mHealth app to their smartphones and complete the intervention within 6 weeks. They will be required to complete daily electronic sleep diaries for the following 6 weeks. Each week, they will be asked to complete a short assessment of their experiences from the previous week and their current insomnia severity
  Arms: mHealth application
Device: Simplified mHealth application and sleep health education — Study participants will download the mHealth app to their smartphones and complete the intervention within 6 weeks. They will receive a simplified version of the app with sleep hygiene instructions and will be required to complete daily electronic sleep diaries for the following 6 weeks. Each week, they will be asked to complete a short assessment of their experiences from the previous week and their current insomnia severity.
  Arms: Control Group

SUMMARY:
This study is to develop and test a medical health application based on cognitive behavioral therapy for insomnia and augmented with other evidence-based sleep interventions that address common sleep-related problems in opioid use disorder. An initial program will be built utilizing input from persons beginning medications for opioid use disorders.

DETAILED DESCRIPTION:
This pilot randomized controlled trial will assess the feasibility and acceptability of an evidence-based behavioral sleep intervention delivered via a mHealth app to individuals initiating treatment with medications for opioid use disorder. Additional outcomes include changes in sleep disturbance over the course of the 6-week intervention. Participants (N=40, 20 per group) will be randomized to download the mHealth app to their smartphones and complete the intervention within 6 weeks. The control group will receive a simplified version of the app with sleep hygiene instructions. Both groups will complete daily electronic sleep diaries for the following 6 weeks. Each week, they will be asked to complete a short assessment of their experiences from the previous week and their current insomnia severity. At the end of the 6th week, they will complete an online series of questionnaires, including validated feasibility/acceptability measures and measures of insomnia severity.

ELIGIBILITY:
Inclusion Criteria:

* No experience of withdrawal symptoms in past 2 weeks
* Being stabilized on buprenorphine

  1. Initiated buprenorphine in past 3 months
  2. Modified buprenorphine dose in past 3 months (e.g., reducing dose with goal of transitioning to vivitrol)
* Currently experiencing clinically significant sleep disturbance (PSQI > 5)
* Able to read and understand English
* Owns an Android or iOS smartphone
* At least 18 years of age

Exclusion Criteria:

* Current psychotic symptoms
* Current active suicidal ideation
* Severe visual impairment
* Current use of benzodiazepines
* Current severe SUD other than OUD (i.e., > 5 criteria met for any other SUD type per DSM-5)
* Peripartum women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Enrollment feasibility/acceptability benchmark of at least 30 persons completing entire study period - Enrollment and retention percentages | 6 weeks following enrollment
  To achieve a minimum enrollment and retention percentage of 75% throughout the 6-week investigation period.
Protocol adherence feasibility/acceptability benchmarks of participants completing modules and sleep diaries each week - Engagement | 6 weeks following enrollment
  Completing at least one module per week, submitting a minimum of four sleep diaries per week, and implementing stimulus control and sleep restriction on at least 90% of nights.
mHealth App Usability Questionnaire | 6 weeks following enrollment
  Validated measure of mobile app usability with 3 sections: Ease of use/satisfaction, system information arrangement, and usefulness

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | At enrollment and 6 weeks following enrollment
  Validated measure of difficulty falling and staying asleep and subsequent daytime function
Structured Clinical Interview for Sleep Disorders - Revised Edition | At enrollment and 6 weeks following enrollment
  Assessment for sleep disorders based on the DSM-5
Insomnia Severity Index | At enrollment and 6 weeks following enrollment
  Global sleep quality; the most common self-reported sleep measure
Daily Sleep Diary - Sleep Onset Latency | Through study completion of 6 weeks
  Subjective sleep onset latency (time to fall asleep)
Daily Sleep Diary - Wake-time After Sleep | Through study completion of 6 weeks
  Subjective time awake after sleep onset
Daily Sleep Diary - Total Sleep Time | Through study completion of 6 weeks
  Subjective total sleep time
Daily Sleep Diary - Sleep Efficiency | Through study completion of 6 weeks
  Subjective sleep efficiency

OTHER OUTCOMES:
MOUD and drug use | Through study completion of 6 weeks
  Self-reported checklist

CONTACTS AND LOCATIONS:
Overall Officials: Allison K Wilkerson, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No